CLINICAL TRIAL: NCT06099210
Title: The Value of Multimodal MR Imaging in Cognitive Assessment of Patients With Moderate Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Ankang Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-194
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Brain Injuries
Keywords: moderate traumatic brain injury; MRI; axial cord injury; cognitive disorder
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate traumatic brain injury: Intervention: Glasgow coma scale
  Interventions: Diagnostic Test: Glasgow coma scale
- Healthy control group

INTERVENTIONS:
Diagnostic Test: Glasgow coma scale — Closed tach brain injury due to external force was included according to the GCS score
  Groups: Moderate traumatic brain injury

SUMMARY:
The goal of this observational study is to learn about in The value of multimodal MR Imaging in cognitive assessment of patients with moderate traumatic brain injury. The main question it aims to answer is:

• The construction of the core injury model of cognitive impairment caused by moderate brain trauma takes multi-parameter MR scanning as the main line of research, centering on the analysis of cognitive impairment of white matter structure damage and brain function involved in the research institute, and conducts research on key scientific issues such as the validity verification of cognitive prognosis after moderate brain trauma.

Participants will be collected for MR, hematology and stool and neuropsychological Scale indicators in the study.

DETAILED DESCRIPTION:
According to the World Health Organization's (WHO) public health statistics on neurological diseases, it is expected that by 2030, neurological injuries caused by brain trauma will become the leading cause of disability of neurological diseases, and Alzheimer's disease and cerebrovascular disease combined two to three times. More than 50 million people worldwide suffer from TBI each year, and about half of the world's population may experience one or more TBI in their lifetime. As a potential risk factor, TBI will increase the risk of neurodegenerative diseases by 1.5 times, and up to 30%-70% of TBI patients will develop neurological symptoms. Brain injury is an important global medical, public health and social problem. Early diagnosis and effective treatment can effectively reduce the disability rate of patients and the incidence of neurological sequelae, which has become a hot topic in the international scientific research community. This study focuses on the construction of the core injury model of cognitive impairment caused by moderate traumatic brain injury, takes multi-parameter MR Scanning as the main line of research, and focuses on the analysis of cognitive impairment caused by white matter structure injury and brain function covariation involved in this study as the breakthrough point, and carries out research on key scientific issues such as the validity verification of cognitive prognosis after moderate traumatic brain injury.

This study was conducted mainly on moderate brain trauma, combined with related departments of neurosurgery, imaging, laboratory, rehabilitation and pain. The research objective is to collect 50 patients with brain trauma and 50 healthy control group from the First Affiliated Hospital of Xi'an Jiaotong University and Ankang Central Hospital. The magnetic resonance, hematology, stool and neuropsychology scale 3 indicators. Magnetic resonance examination: For patients with moderate craniocerebral trauma who meet the inclusion criteria, head MRI scans were performed in the subacute period after injury (within 10 to 21 days) and 3-6 months (chronic phase); for the control group with age, gender, education, skill and disease group and with no psychiatric or neurological diseases. The scanning sequence includes: (1) 3-pl (the positioning image requires the preservation of the whole brain, Including the overhead scalp to all the cerebellum) (check the parameters before scanning); (2) T2-FLAIR (brain condition prediction, If any abnormal lesion, The scan should be stopped immediately) (3) T1-weighted 3D-MPRAGE (4) DTI (5) Resting State (BOLD) (positioning line parallel to AC-PC line) (6) MAGiC (7) ASL 5. Neuropsychological evaluation: patients with moderate brain trauma before or within 48 hours after each scan; For healthy controls matched for sex, age, education, and literacy, Neuropsychological scale assessments were performed at 48 hours after completing the MRI examination. The scale includes pain after TBI, memory, executive function, information processing, TBI recovery, anxiety, and depression.6. Hematology and stool data collection: collect data of hematological markers (whole blood samples to our hospital (0 days), the first MR scan (10~21 days) and 24 hours before (3-6 months after injury) (3 mL * 2, serum samples 3 mL * 1 / time), collect stool samples (about 1mg) before the first MR scan and 24 hours before the second MR scan.

ELIGIBILITY:
Inclusion Criteria:

* GCS 9-12 points
* Time for loss of consciousness: 30 minutes-24 hours
* Forget time after injury: 1-7 days

Exclusion Criteria:

* Alcohol consumption, substance abuse during or within the previous 24 hours
* Previous history of traumatic brain injury, MRI contraindication, penetrating brain injury, psychotropic substance use, spinal cord injury, positive neurological examination, multifunctional disorder
* Neurological and psychiatric history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Inclusion criteria: emergency admission. Age: 18-60 years, GCS 9-12 points at presentation, time for loss of consciousness: 30 minutes-24 hours, forgetting time after injury: 1-7 days.2. Control group: in the age, gender, education level, skill and disease group matching, and no psychiatric or neurological diseases.3. Exclusion criteria: alcohol consumption within 24 hours at the time or before, and drug abuse. Previous history of brain trauma, MRI contraindication, brain penetrating injury, psychotropic drug use, spinal cord injury, positive neurological examination, multifunctional disorder, neurological and psychiatric history with significant MRI artifacts, and poor image quality.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
head MRI scans | in the subacute period after injury (within 10 to 21 days) and 3-6 months (chronic phase)
  The scanning sequence includes: (1) 3-pl (the positioning image requires the preservation of the whole brain, Including the overhead scalp to all the cerebellum) (check the parameters before scanning); (2) T2-FLAIR (brain condition prediction, If any abnormal lesion, The scan should be stopped immediately) (3) T1-weighted 3D-MPRAGE (4) DTI (5) Resting State (BOLD) (positioning line parallel to AC-PC line) (6) MAGiC (7) ASL
Neuropsychological evaluation | patients with moderate brain trauma before or within 48 hours after each scan; For healthy controls matched for sex, age, education, and literacy, Neuropsychological scale assessments were performed at 48 hours after completing the MRI examination.
  The scale includes pain after TBI, memory, executive function, information processing, TBI recovery, anxiety, and depression.
  Questionnaires were scored separately. Trail making test A: The score is given in time (seconds). If the test time is greater than 78 seconds, the higher the score, the worse the damage is. Rivermead Post Concussion: From 0 to 80, the higher the score may reflect the more severe the sequelae of concussion. Digit Span: From 0-12, higher scores may reflect better number breadth. Language fluency test: greater than or equal to 0 points, the higher the score, the better the language fluency. Pain score: 0-50, the higher the score reflects the higher pain. Short From Headache Impact Test: 36-78 points, higher scores reflect higher headache degree. Fatigue Severity Scale: 1-7, and higher scores reflect greater fatigue. Mini-mental State Examination: Less than or equal to 22 is dementia, and less than or equal to 15 is severe dementia.
Hematology and stool data | hematological markers (whole blood samples (0 days), the first MR scan (10~21 days) and 24 hours before (3-6 months after injury), stool samples before the first MR scan and 24 hours before the second MR scan.)
  collect data of hematological markers (whole blood samples to our hospital (0 days), the first MR scan (10~21 days) and 24 hours before (3-6 months after injury) (3 mL * 2, serum samples 3 mL * 1 / time), collect stool samples (about 1mg) before the first MR scan and 24 hours before the second MR scan.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No